CLINICAL TRIAL: NCT04092634
Title: Dual-mobility vs. Single-bearing Components in THA at "High Risk" for Prosthetic Dislocation
Brief Title: Dual Mobility in "High Risk" Patients
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: New York University (Other); Rothman Institute Orthopaedics (Other); Keck School of Medicine of USC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17030101
Record Dates: First submitted 2019-09-11; First posted 2019-09-17 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Dislocation, Hip
MeSH Terms: conditions — Hip Dislocation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two groups: THA with dual mobility components vs THA with single-bearing designs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Dual mobility (Experimental): Patients in this group will receive a dual mobility hip implant
  Interventions: Device: Dual mobility implant
- Single bearing, traditional hip implant (Active Comparator): Patients in this group will receive a traditional, single-bearing hip implant.
  Interventions: Device: Traditional, Single-bearing hip implant

INTERVENTIONS:
Device: Dual mobility implant — Patients that are eligible and consent to the study will be randomized to receive either a dual mobility implant or a traditional single-bearing hip implant. This group is for the dual mobility implant
  Arms: Dual mobility
Device: Traditional, Single-bearing hip implant — Patients that are eligible and consent to the study will be randomized to receive either a dual mobility implant or a traditional single-bearing hip implant. This group is for the dual mobility implant
  Arms: Single bearing, traditional hip implant

SUMMARY:
The aim of this study is to compare clinical outcomes of patients considered to be high risk for prosthetic dislocation undergoing primary total hip arthroplasty (THA) with the use of a dual mobility bearing versus a conventional, single bearing design.

DETAILED DESCRIPTION:
This study aims to compare the clinical outcomes of patients considered to be at high risk for prosthetic dislocation undergoing primary total hip arthroplasty (THA) with the use of a dual mobility bearing versus a conventional, single-bearing design.

We hypothesize that in primary THA patients considered to be at high risk for prosthetic dislocation, the use of dual-mobility components will be associated with a lower dislocation rate in the first year following the index procedure. We do not anticipate a difference. In other clinical outcome measures or functional outcome scores between the two cohorts.

Study Design: Randomized controlled trial with two groups: THA with dual mobility.

44 components vs THA with single-bearing designs

ELIGIBILITY:
Inclusion Criteria:

* Primary THA for a diagnosis of osteoarthritis or inflammatory arthritis in the setting of a history of prior lumbar or lumbosacral fusion performed at least 6 months prior to their THA. In addition, patients considered high-risk for potential prosthetic dislocation will be included based on the presence of one or more of the following: neuromuscular disorder (e.g. cerebral palsy, Parkinson's disease, history of a stroke), dementia or cognitive impairment, substance or alcohol abuse (>10 drinks per week), acute displaced femoral neck fracture, age > 75 years, inflammatory arthritis, and increased preoperative range of motion (calculated as described by Krenzel et al.: combined flexion, adduction, internal rotation > 115 degrees).

Exclusion Criteria:

* Less than 18 years of age
* Revision THA
* spinopelvic fusion that is more recent than 6 months prior to THA
* isolated cervical or thoracic fusion
* intent to undergo a revision spinopelvic fusion within one year of their index THA
* a history of prior infection in the affected hip
* a history of prior open surgery on the affected hip (i.e. prior proximal femur fracture or osteotomy)
* or a preoperative diagnosis of post-traumatic arthritis, avascular necrosis, or fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2035-02-01 (Estimated)

PRIMARY OUTCOMES:
Hip Dislocation | 6 weeks following their index surgical procedure.
  The rate of prosthetic dislocation between the two cohorts
Hip Dislocation | 1 year following their index surgical procedure.
  The rate of prosthetic dislocation between the two cohorts
Hip Dislocation | 2 years following their index surgical procedure.
  The rate of prosthetic dislocation between the two cohorts
Hip Dislocation | 5 years following their index surgical procedure.
  The rate of prosthetic dislocation between the two cohorts
Hip Dislocation | 10 years following their index surgical procedure.
  The rate of prosthetic dislocation between the two cohorts

SECONDARY OUTCOMES:
Complications | Complications will be assess up to 10 years following their index surgical procedure
  Any peri- or postoperative complications will be recorded component loosening, occurrence of intraprosthetic dislocation, infection, periprosthetic fractures, revision rates
Radiographic signs of loosening and proper component placement. | 6 weeks following their index surgical procedure.
  Routine radiographs (AP Pelvis, frogleg lateral, and cross-table lateral radiographs) will be obtained at follow-up visits and assessed for cup placement, anteversion, radiographic signs of loosening, and component migration. These radiographs will be assess for the presence of loosening in a yes/no format
Radiographic signs of loosening and proper component placement. | 1 year following their index surgical procedure.
  Routine radiographs (AP Pelvis, frogleg lateral, and cross-table lateral radiographs) will be obtained at follow-up visits and assessed for cup placement, anteversion, radiographic signs of loosening, and component migration. These radiographs will be assess for the presence of loosening in a yes/no format
Radiographic signs of loosening and proper component placement. | 2 years following their index surgical procedure.
  Routine radiographs (AP Pelvis, frogleg lateral, and cross-table lateral radiographs) will be obtained at follow-up visits and assessed for cup placement, anteversion, radiographic signs of loosening, and component migration. These radiographs will be assess for the presence of loosening in a yes/no format
Radiographic signs of loosening and proper component placement. | 5 years following their index surgical procedure.
  Routine radiographs (AP Pelvis, frogleg lateral, and cross-table lateral radiographs) will be obtained at follow-up visits and assessed for cup placement, anteversion, radiographic signs of loosening, and component migration. These radiographs will be assess for the presence of loosening in a yes/no format
Radiographic signs of loosening and proper component placement. | 10 years following their index surgical procedure.
  Routine radiographs (AP Pelvis, frogleg lateral, and cross-table lateral radiographs) will be obtained at follow-up visits and assessed for cup placement, anteversion, radiographic signs of loosening, and component migration. These radiographs will be assess for the presence of loosening in a yes/no format

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Keck School of Medicine of USC, Los Angeles, California
  - Rush University Medical Center, Chicago, Illinois
  - New York University Medical Center, New York, New York
  - Rothman Orthopaedic Institute, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No